CLINICAL TRIAL: NCT05445765
Title: Anti-CD33 CAR-T Cells for the Treatment of Relapsed/Refractory CD33+ Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCar Bio Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG165-001
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Relapsed and/or Refractory Acute Myeloid Leukemia; High Risk Hematologic Malignancies
Keywords: CD33; anti-CD33 CAR; leukemia; acute myeloid leukemia; hematologic malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD33 CAR T cells (Experimental): Dose escalation phase: anti-CD33 CAR T cells will be transduced with a lentiviral vector to express anti-CD33 CARs
  Interventions: Biological: anti-CD33 CAR T cells

INTERVENTIONS:
Biological: anti-CD33 CAR T cells — Anti-CD33 CAR T cells are used to treat patients. Patient will be administered either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of anti-CD33 CAR-T cells in patients with relapsed and/or refractory, high risk hematologic malignancies.

DETAILED DESCRIPTION:
AML is a rapidly progressing blood cancer and treated by high-dose multi-agent chemotherapy potentially followed by hematopoietic stem cell transplantation. Despite such intensive therapies, which are often associated with considerable toxicities and even death, about 60-70% of AML patients still relapse. Furthermore, the five-year survival rate from AML remains at a dismal 27%. AML is composed mostly of CD33+ leukemic blast cells. Therefore, CD33 is a potential good target by CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent; Patients volunteer to participate in the clinical trial;
2. Diagnosis is mainly based on the World Health Organization (WHO) 2008;
3. Complete remission cannot be achieved after induction therapy; recurrence occurs after completion remission; the burden of leukemic blasts in the peripheral blood or bone marrow is greater than 5%;
4. Leukemic blast cells express CD33 (CD33 positive by flow cytometry or immunohistochemistry ≥70%);
5. The expected survival period is greater than 12 weeks;
6. ECOG score ≤2;
7. Age 2-60 years old;
8. HGB≥70g/L (can be transfused);
9. Total bilirubin does not exceed 3 times the upper limit of normal value, and AST and ALT do not exceed 5 times the upper limit of normal value.

Exclusion Criteria:

1. Patients declining to consent for treatment
2. Prior solid organ transplantation
3. One of the following cardiac issues: atrial fibrillation; myocardial infarction within the past 12 months; prolonged QT syndrome or secondary QT prolongation; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV;
4. History of severe pulmonary dysfunction diseases;
5. Severe infection or persistent infection cannot be effectively controlled;
6. Severe autoimmune disease or congenital immunodeficiency;
7. Active hepatitis;
8. Human immunodeficiency virus (HIV) infection;
9. Clinically significant viral infections, or uncontrollable viral reactivation, including EBV (Epstein-Barr virus).

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The number and incidence of adverse events after anti-CD33 CAR infusion. | 1 year, particularly the first 3 months after CAR infusion
  Determine the toxicity profile of anti-CD33 CAR T cell therapy including the number, incidence, and severity of symptoms such as cytokine release syndromes and neurotoxicity

SECONDARY OUTCOMES:
The disease response to anti-CD33 CAR T cells | 4 weeks
  The disease response to anti-CD33 CAR T cells is evaluated by bone marrow biopsy and aspirate at 1, 2, 3, and 4 weeks. The proportion of subjects receiving anti-CD33 CAR T infusion to 1) morphological remission (blasts <5%): 2) flow cytometry analysis was blast negative, and 3) molecular biological remission (if applicable).
Allogeneic hematopoietic stem cell transplantation (HCT) | 42 days after HCT ingraftment
  Allogeneic hematopoietic stem cell transplantation (HCT) is performed after anti-CD33 CAR T treatment. The time after HCT engraftment [time range: 42 days after HCT ingraftemnt] is calculated from the day of HCT until the absolute neutrophil count (ANC) is greater than 500 / ul for three consecutive days.
HCT 100% chymerism time | 2 weeks after HCT
  HCT 100% chymerism time
Overall survival | 1 year after HCT
  The time from the start of anti-CD33 CAR T injection to death is determined as the overall survival
Progress-free survival | one year after HCT
  Progress-free survival is measured from the injection of anti-CD33 CAR T cells until the record of disease progression or death due to any reason, whichever comes first.
Treatment-related mortality | one year after HCT
  Treatment-related mortality calculated from one year after HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD, Principal Investigator — Hebei Yanda Lu Daopei Hospital
Locations (1):
- Hebei Yanda Lu Daopei Hospital, Langfang, Hebei, China